CLINICAL TRIAL: NCT00351377
Title: Measurement and Analysis of Patient Reported Gastrointestinal (GI) and Health-related Quality of Life (HRQL) Outcomes in Patients With Autoimmune Diseases Treated With Mycophenolate (MPA)
Brief Title: Gastrointestinal and Health-related Quality of Life Outcomes in Patients With Autoimmune Diseases Treated With Mycophenolate
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CERL080ADE08
Record Dates: First submitted 2006-07-10; First posted 2006-07-12 (Estimated); Results first posted 2011-01-12 (Estimated); Last update posted 2011-04-21 (Estimated); Status verified 2011-04

CONDITIONS: Autoimmune Disease
Keywords: Autoimmune disease, mycophenolate, GI problems
MeSH Terms: conditions — Autoimmune Diseases | interventions — Mycophenolic Acid

ARMS (1):
- Enteric-coated Mycophenolate Sodium (Experimental): Enteric-coated Mycophenolate Sodium (EC-MPS) 180 mg and 360 mg tablets were administered orally in divided doses twice daily in a dose that was equimolar to the dose of Mycophenolate mofetil the participant was taking at the time of study entry. The planned duration of treatment 6 to 8 weeks.
  Interventions: Drug: Enteric-coated Mycophenolate Sodium

INTERVENTIONS:
Drug: Enteric-coated Mycophenolate Sodium — Enteric-coated Mycophenolate Sodium (EC-MPS) 180 mg and 360 mg tablets were administered orally in divided doses twice daily.
  Other Names: Myfortic

SUMMARY:
Treatment with the immunosuppressive drug mycophenolate mofetil (MMF) may result in gastrointestinal (GI) complications in some patients. This study will 1) determine the proportion of patients with autoimmune diseases who are experiencing any GI complaints under MMF-based immunosuppressive treatment and 2) assess if a switch from MMF to enteric-coated mycophenolate sodium (EC-MPS) results in improved GI and/or health-related quality of life outcomes.

ELIGIBILITY:
Inclusion criteria:

1. Patients with autoimmune diseases;
2. receiving immunosuppressive therapy that includes MMF at time of study enrollment;
3. receiving immunosuppressive regimen that includes MMF at a stable dose for at least 1 month prior to enrollment. Patients can only be enrolled into the study if it is expected that treatment will continue at the same dose until study end (6-8 weeks after enrollment).

Exclusion criteria:

1. If applicable, GI symptoms assumed or known not to be caused by Mycophenolic acid (MPA) therapy (e.g. oral biphosphonates induced, infectious diarrhea);
2. Women of child-bearing potential who are planning to become pregnant or are pregnant and/or lactating or who are unwilling to use effective means of contraception;
3. Presence of psychiatric illness (i.e., schizophrenia, major depression) that, in the opinion of the site investigator, would interfere with study requirements;
4. Current acute medical intervention or hospitalization;
5. Presence of a medical condition not related to a GI event at time of visit, which requires immediate medical intervention.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2006-06; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigational Site, Various Cities, Germany

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Enteric-coated Mycophenolate Sodium
Started | 111
Completed | 104
Not Completed | 7
Not completed — Adverse Event | 5
Not completed — Death | 1
Not completed — Unsatisfactory therapeutic effect | 1

BASELINE CHARACTERISTICS:
Arm/Group | Enteric-coated Mycophenolate Sodium
Number analyzed (Participants) | 111
Age Continuous [Mean (Standard Deviation); unit: years] | 49.5 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82
  Male | 29

OUTCOME MEASURES:

1. Primary Outcome: Changes in GI Symptom Severity After Conversion From Mycophenolate Mofetil (MMF) to Enteric-coated Mycophenolate Sodium (EC-MPS)
Description: Changes in GI symptom severity was measured by changes in the Gastrointestinal Symptom Rating Scale (GSRS) total score from baseline visit to the visit at 6-8 weeks. This total score was calculated as the average of the 15 single items (each ranging from 1-7 score points) and thus also had a range from 1-7 score points. Higher values indicate more unfavorable conditions.
Time Frame: Baseline and 6 - 8 weeks
Population: Intention to treat (ITT) population consisting of all enrolled participants who received study medication.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Enteric-coated Mycophenolate Sodium
Number analyzed (Participants) | 111
Scores on a scale
  Baseline (N= 111) | 2.28 (1.13)
  6-8 Weeks (N= 102) | 2.02 (0.93)
  Change From Baseline (N = 102) | -0.28 (0.92)

2. Secondary Outcome: Changes in the GI Symptom Severity Subscales After Conversion to Enteric-coated Mycophenolate Sodium
Description: Changes in GI symptom severity was measured by changes in the total scores of 5 subscales (reflux, diarrhea, constipation, abdominal pain and indigestion) of the Gastrointestinal Symptom Rating Scale (GSRS) from baseline visit to the visit at 6-8 weeks. The GSRS is a 15-item instrument with a mean subscale score ranging from 1 (no discomfort) to 7 (very severe discomfort).
Time Frame: Baseline and 6-8 weeks
Population: Intention to treat (ITT) population consisting of all enrolled participants who received study medication.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Enteric-coated Mycophenolate Sodium
Number analyzed (Participants) | 111
Scores on a scale
  Reflux [n =102] | -0.24 (1.36)
  Diarrhea [n =104] | -0.27 (1.43)
  Constipation [n = 104] | 0.02 (1.18)
  Abdominal pain [n =102] | -0.51 (1.20)
  Indigestion [n = 104] | -0.42 (1.33)

3. Secondary Outcome: Changes in GI-related Quality of Life Index (GIQLI), After Patients Are Converted From MMF to Enteric-coated Mycophenolate Sodium
Description: Assessed by changes in the Gastrointestinal Quality of Life Index (GIQLI) from Baseline visit to the 6-8 week visit. The GIQLI is a 36-item questionnaire and consists of 5 different subscales. The total score was calculated as the sum of the 36 single items which each ranged from 0-4, leading to a hypothetical range from 0-144 score points (lower scores indicate more unfavorable conditions). The mean change was calculated as (6-8 week visit value) minus (Baseline value).
Time Frame: Baseline and 6-8 weeks
Population: Intention to treat (ITT) population consisting of all enrolled participants who received study medication.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Enteric-coated Mycophenolate Sodium
Number analyzed (Participants) | 111
Scores on a scale
  Baseline (N= 111) | 100.2 (23.8)
  6-8 Weeks (N= 104) | 105.6 (22.9)
  Change from Baseline (N= 104) | 5.8 (18.6)

4. Secondary Outcome: Changes in the GI-related Quality of Life Subscales After Conversion to Enteric-coated Mycophenolate Sodium
Description: The 5 different subscales of the GI-related Quality of Life (GIQLI) were analyzed separately by calculating the average value of the items that were included in the respective subscore. Thus, the theoretical range for each of the subscores was the same as for the single items, i.e. 0-4 score points. An increase in the subscale score indicates an improvement in symptoms.
Time Frame: Baseline and 6-8 weeks
Population: Intention to treat (ITT) population consisting of all enrolled participants who received study medication.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Enteric-coated Mycophenolate Sodium
Number analyzed (Participants) | 111
Scores on a scale
  GI symptoms [n=103] | 0.18 (0.53)
  Emotional status [n=103] | 0.15 (0.68)
  Physical function [n=102] | 0.22 (0.68)
  Social function [n=102] | 0.10 (0.66)
  Stress of medical treatment [n=102] | 0.19 (1.22)

5. Secondary Outcome: Changes in Psychological General Well-Being Index (PGWB) After Conversion to Enteric-coated Mycophenolate Sodium
Description: The PGWB consists of 22 single items (each ranging from 0-5) with 7 dimensions (including the total score) to be calculated. Lower scores indicate more unfavorable conditions. The total raw score is calculated by summing up all of the single items and thus has a hypothetical range from 0-110 score points. This raw score is further transformed using the formula: (raw score / 110) x 100 to fit a range from 0-100.
Time Frame: Baseline and 6-8 weeks
Population: Intention to treat (ITT) population consisting of all enrolled participants who received study medication.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Enteric-coated Mycophenolate Sodium
Number analyzed (Participants) | 110
Scores on a scale
  Baseline (N= 110) | 65.3 (16.1)
  6-8 Weeks (N= 103) | 66.8 (15.6)
  Change From Baseline (N= 103) | 2.0 (11.1)

6. Secondary Outcome: Changes in Psychological General Well-Being Index (PGWB) Subscales After Conversion to Enteric-coated Mycophenolate Sodium
Description: The change from baseline to the 6-8 week visit for each of the six subscores (each ranging from 0-5) of the PGWB were analyzed individually. Each of the subscores was transformed to fit a range from 0-100. Lower scores indicate more unfavorable conditions, so an increase in score indicates an improvement in symptoms.
Time Frame: Baseline and 6-8 weeks
Population: Intention to treat (ITT) population consisting of all enrolled participants who received study medication.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Enteric-coated Mycophenolate Sodium
Number analyzed (Participants) | 111
Scores on a scale
  Anxiety [n=103] | 1.3 (14.1)
  Depressed mood [n=104] | 1.5 (14.1)
  Positive well-being [n=104] | 0.7 (14.4)
  Self control [n=104] | 1.5 (15.0)
  General health [n=104] | 3.4 (15.1)
  Vitality [n=104] | 2.7 (16.0)

7. Secondary Outcome: Overall Treatment Effects for GI Symptoms Assessed by the Physician
Description: Assessed using the Overall Treatment Effects for GI symptoms questionnaire. The question was: "Has there been any change in the participant's GI symptoms since his/her last study visit? Please indicate if there has been any change in his/her symptoms." The possible answers were: "Improved", "about the same", or "worse. The questionnaire was completed by the physician.
Time Frame: 6-8 week
Population: Intention to treat population consisting of all enrolled participants who received study medication.
Measure: Number; unit: Participants
Arm/Group | Enteric-coated Mycophenolate Sodium
Number analyzed (Participants) | 111
Participants
  Improved | 49
  About the same | 43
  Worsened | 13
  Missing data | 6

8. Secondary Outcome: Overall Treatment Effects for GI Symptoms Assessed by the Patient
Description: Assessed using the Overall Treatment Effects for GI symptoms questionnaire. The question was: "Has there been any change in the participant's GI symptoms since his/her last study visit? Please indicate if there has been any change in his/her symptoms." The possible answers were: "Improved", "about the same", or "worse. The questionnaire was completed by the patient.
Time Frame: 6-8 week
Population: Intention to treat population consisting of all enrolled participants who received study medication.
Measure: Number; unit: Participants
Arm/Group | Enteric-coated Mycophenolate Sodium
Number analyzed (Participants) | 111
Participants
  Improved | 38
  About the same | 53
  Worsened | 9
  Missing data | 11

9. Secondary Outcome: Overall Treatment Effects for for Health-related Quality of Life Assessed by the Patient
Description: Assessed using the Overall Treatment Effects for health-related quality of life questionnaire. Possible answers were: "Improved", "about the same", or "worse. The questionnaire was completed by the patient.
Time Frame: 6-8 week
Population: Intention to treat population consisting of all enrolled participants who received study medication.
Measure: Number; unit: Participants
Arm/Group | Enteric-coated Mycophenolate Sodium
Number analyzed (Participants) | 111
Participants
  Improved | 31
  About the same | 61
  Worsened | 10
  Missing data | 9

ADVERSE EVENTS:
Arm/Group | Enteric-coated Mycophenolate Sodium
Serious Adverse Events (participants affected / at risk) | 6/111
Other Adverse Events (participants affected / at risk) | 38/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enteric-coated Mycophenolate Sodium (N=111)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Diverticulum (Gastrointestinal disorders) | 1
Bronchitis (Infections and infestations) | 1
Endocarditis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Dementia (Nervous system disorders) | 1
Disturbance in attention (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Enteric-coated Mycophenolate Sodium (N=111)
Abdominal distension (Gastrointestinal disorders) | 8
Diarrhoea (Gastrointestinal disorders) | 16
Dyspepsia (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 13
Vomiting (Gastrointestinal disorders) | 10
Nasopharyngitis (Infections and infestations) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.